CLINICAL TRIAL: NCT01283568
Title: Phase IV Study of Combined GAMALINE and HIPERICIN for Treating Pre-Menstrual Syndrome and Vasomotor Symptoms
Brief Title: Safety and Efficacy Study of Gamaline+Hipericin in PMS
Acronym: GH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Phytopharm Consulting Brazil (Network)
Collaborators: Herbarium Laboratorio Botanico Ltda (Industry); Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: GAMALINEHIPERICIN
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Edema; Depression; Hot Flashes; Anxiety; Irritability
Keywords: PMS, climacteric, depression
MeSH Terms: conditions — Edema; Depression; Hot Flashes; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1 - Gamaline+Hipericin - fertile women
- 2- Gamaline+Hipericin - climateric women
- 3- Gamaline- control - fertile women
- 4 - Gamaline control - climateric women

SUMMARY:
GAMALINE is already register for PMS and HIPERICIN as antidepressive drug. Both plant extracts. The investigators will try the mixture and see if the vasomotor symptoms will disappear. The investigators expect that together all symptoms will be covered better than Gamaline alone. The investigators will run for 180 days measuring at T0, T1 and T6 (starting point, 30 days and 180 days).

DETAILED DESCRIPTION:
This protocol wants to show the advantages for the mixture GAMALINE 900mg+HIPERICIN 300mg - 2 herbal extracts for PMS treatment against the individual use of GAMALINE

ELIGIBILITY:
Inclusion Criteria:

* climacteric pre-menopausal women between 45 e 55 anos
* women between 25 e 44 anos

Exclusion Criteria:

* Age inferior 25 anos or superior 55 anos and/or decline invitation.
* Patients pos-menopause
* Under hormone therapy
* Thyroid disease
* Under psychiatric therapy or medication
* History for allergies and hypersensitivity to one or both extracts
* Breast feeding or pregnancy
* No knowledge for writing and/or reading

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Only women from 25 to 55 years old with PMS symptoms
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Karla F Deud José, Pharm PhD, Study Chair — Phytopharm Consulting Brazil - karla@phytopharm.com.br
Locations (1):
- Ambulatório de Ginecologia e Obstetrícia ISCMPA, Porto Alegre, Rio Grande do Sul, Brazil